CLINICAL TRIAL: NCT06612489
Title: Efficacy of Biofeedback-Based Serious Game for Pain Alleviation in Middle-Aged and Older Ovarian Cancer Patients: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Jianan Zhao, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: biofeedback based game
Record Dates: First submitted 2024-06-13; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: The intervention product consists of a serious game designed to facilitate digitalized distraction therapy, integrated with a wearable device that monitors the user's real-time immersion level. The serious game is presented as a mobile game where users must consistently identify target elements following a specific rhythm to achieve a distraction effect. The game theme, centered around fishing and music, was chosen to align with the hobbies of the target population. Design elements were carefully selected based on age-friendly design criteria from previous research.The wearable device features the TGAM chip as its central component, which captures electroencephalogram (EEG) signals from the patients and processes them to derive an immersion level score.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention consist of 26 participants using biofeedback based dynamic-difficulty game for 15 mins each.
  Interventions: Device: biofeedback based dynamic-difficulty game
- Control group (Other): Twenty six participants in the control group played a serious game with a fixed difficulty level for 15 mins each
  Interventions: Device: fixed difficulty game

INTERVENTIONS:
Device: biofeedback based dynamic-difficulty game — A biofeedback based dynamic-difficulty serious game rooted in distraction therapy.
  Arms: Intervention group
Device: fixed difficulty game — A fixed difficulty serious game rooted in distraction therapy.
  Arms: Control group

SUMMARY:
Consistent pain affects most middle-aged and older ovarian cancer patients. Non-pharmacological pain interventions, such as serious games, offer a promising approach to alleviating this pain by providing an effective sense of immersion. However, current games on the pain alleviation lack examination of its efficacy in middle-aged and older population and real-time monitoring of immersion level, particular since immersion level is highly associated with pain alleviation effect and adjustable to challenging level of game difficulty. This study developed a serious game with biofeedback-driven dynamic difficulty. Then examined its feasibility and efficacy through a two-arm, single-blinded randomized controlled trial. A total of 52 participants were recruited and randomized into intervention group and control group to receive biofeedback-based dynamic-difficulty serious game or fix-difficulty serious game for 15 mins each, respectively. The primary outcome was the assessment of the pain level, measured using the Visual Analog Scale. The secondary outcomes included pain-related anxiety, immersion level, and user experience.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic standards established by the International Association for the Study of Pain (IASP) and having a pain severity level between 3 and 6 (classified as mild to moderate) at the time of enrollment,
* Diagnosed with ovarian caner
* Demonstrating clear cognitive and expressive abilities,
* Being aged 45 or older,
* Providing voluntary consent after fully understanding the study's objectives.

Exclusion Criteria:

* Individuals with a history of mental illness or communication disorders,
* Those experiencing vision or cognitive impairments,
* Individuals undergoing pain medication treatment during the intervention period.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Pain level | 15 mins
  Patients' pain perception was assessed using the Visual Analog Scale (VAS), a widely accepted tool in clinical settings due to its convenience and ease of understanding. The VAS employs a 10-scale ruler from 1 to 10 with a movable marker, where higher number indicating a more severe level of pain. Patients are instructed to place the marker on the ruler at the point that corresponds to their current level of pain.

SECONDARY OUTCOMES:
Pain related anxiety | 15 mins
  The Psychological Assessment of the Symptoms of Pain (PASS) scale was used to evaluate patients' psychological states during painful episodes. This scale consists of four subscales - cognition, avoidance, fear, and physiological anxiety - each containing five items, totaling 20 items. Responses are rated on a 5-point Likert scale from 0 to 4, with higher scores indicating greater levels of pain-related anxiety and fear. The PASS scale demonstrates good reliability and validity, providing a scientific means of assessing pain-related psychological distress.
Immersion level | 15 mins
  Immersion level was assessed using a combination of objective and subjective measures. Physiological data on immersion level indicators were obtained through the wearable EEG device using the TGAM brainwave monitoring module, while subjective evaluation was conducted using the Attention Control Scale (ACS). The ACS comprises two subscales: Attention Focus and Attention Shift. This study utilized the Attention Shift subscale to measure improvements in patients' ability to shift attention after intervention. Each item on the Attention Shift subscale was rated on a Likert scale ranging from 1 to 4, with higher scores denoting more frequent occurrences, thus shedding light on patients' attentional control capabilities and their aptitude to redirect focus.

OTHER OUTCOMES:
User experience | 15 mins
  The user experience of the game was evaluated using the short version of the User Experience Questionnaire (UEQ-S). Participants provided ratings for each item on a 7-point scale, from -3 (negative) to 3 (positive). Higher scores on each scale indicated a more favorable user experience in that dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Jianan Zhao, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable requests.